CLINICAL TRIAL: NCT00540995
Title: Phase I/II Study of Intravenous (IV) Busulfan and Etoposide (VP-16) Combined With Escalated Doses of Large Field Image-Guided Intensity Modulated Radiation Therapy (IMRT) Using Helical Tomotherapy as a Preparative Regimen for Allogeneic Hematopoietic Stem Cell Transplantation (HSCT) for Patients With Advanced Myeloid Malignancies
Brief Title: Busulfan, Etoposide, and Intensity-Modulated Radiation Therapy Followed By Donor Stem Cell Transplant in Treating Patients With Advanced Myeloid Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Unable to safely escalate to TMLI doses that were hypothesized to be effective and less toxic than FTBI. Likely due to the giving of Busulfan prior to radiation delivery. Therefore, the study was abandoned and no further patients were accrued.
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 05013; NCI-2010-00354; CDR0000567452 (Registry Identifier: PDQ)
Record Dates: First submitted 2007-10-05; First posted 2007-10-08 (Estimated); Results first posted 2021-11-22 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Blastic Phase Chronic Myelogenous Leukemia; Childhood Acute Myeloid Leukemia in Remission; Childhood Chronic Myelogenous Leukemia; Childhood Myelodysplastic Syndromes; Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Myeloid Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Refractory Anemia With Excess Blasts
MeSH Terms: conditions — Congenital Abnormalities; Blast Crisis; Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts | interventions — Busulfan; Etoposide; Podophyllotoxin; Radiotherapy, Intensity-Modulated; Transplantation; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I: 1200cGy (Experimental): 1200cGy = 150cGy x 8 doses: Patients receive busulfan IV once daily over 2 hours on days -15 and -13 and then every 6 hours on days -12 to -9. Patients also receive etoposide IV on day -3. Patients undergo image-guided intensity-modulated radiation therapy using helical tomotherapy on days -8 to -5.
  TRANSPLANTATION: Patients undergo allogeneic peripheral blood stem cell transplantation or bone marrow transplantation on day 0.
  GRAFT-VS-HOST DISEASE (GVHD) PROPHYLAXIS: Patients receive GVHD prophylaxis that excludes methotrexate.
  Interventions: Drug: busulfan; Drug: etoposide; Radiation: intensity-modulated radiation therapy; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: allogeneic bone marrow transplantation; Procedure: peripheral blood stem cell transplantation; Radiation: tomotherapy
- Arm II: 1350cGy (Experimental): 1350cGy = 150cGy x 9 doses: Patients receive busulfan IV once daily over 2 hours on days -15 and -13 and then every 6 hours on days -12 to -9. Patients also receive etoposide IV on day -3. Patients undergo image-guided intensity-modulated radiation therapy using helical tomotherapy on days -8 to -5.
  Interventions: Drug: busulfan; Drug: etoposide; Radiation: intensity-modulated radiation therapy; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: allogeneic bone marrow transplantation; Procedure: peripheral blood stem cell transplantation; Radiation: tomotherapy

INTERVENTIONS:
Drug: busulfan — Given IV
  Other Names: BSF; BU; Misulfan; Mitosan; Myeloleukon; Myelosan
Drug: etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; epipodophyllotoxin; VePesid; VP-16; VP-16-213
Radiation: intensity-modulated radiation therapy — Initially 150 cGy X 8 doses with gradual dose escalation to 200 cGy X 10 doses
  Other Names: IMRT
Procedure: allogeneic hematopoietic stem cell transplantation — Stem cell transplantation occurs on Day 0 after High Dose Therapy
Procedure: allogeneic bone marrow transplantation — Stem cell transplantation occurs on Day 0 after High Dose Therapy
  Other Names: bone marrow therapy, allogeneic; bone marrow therapy, allogenic; transplantation, allogeneic bone marrow; transplantation, allogenic bone marrow
Procedure: peripheral blood stem cell transplantation — Stem cell transplantation occurs on Day 0 after High Dose Therapy
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
Radiation: tomotherapy — Initially 150 cGy X 8 doses with gradual dose escalation to 200 cGy X 10 doses
  Other Names: helical tomotherapy

SUMMARY:
RATIONALE: Giving chemotherapy drugs, such as busulfan and etoposide, and intensity-modulated radiation therapy before a donor stem cell transplant helps stop the growth of cancer cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving intensity-modulated radiation therapy together with busulfan and etoposide before a transplant may stop this from happening.

PURPOSE: This phase I/II trial is studying the side effects and best dose of intensity-modulated radiation therapy when given together with busulfan and etoposide followed by a donor stem cell transplant and to see how well it works in treating patients with advanced myeloid cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To establish the maximum tolerated dose (MTD) of a large field image-guided IMRT, using helical tomotherapy, when given in combination with IV busulfan and VP-16 as a preparative regimen for allogeneic hematopoietic stem cell transplantation (HSCT) from an HLA-identical sibling in patients with advanced myeloid malignancies. (Phase I) II. To describe the toxicities at each dose level studied. (Phase I) III. To estimate the radiation doses to the whole body, normal organs, and bone marrow through serial imaging studies following the administration of IMRT. (Phase I) IV. To estimate the overall survival probability, disease-free survival probability, and relapse rate associated with this preparative regimen. (Phase II) V. To characterize the treatment related mortality and toxicity profile (early/late) associated with this regimen. (Phase II) VI. To descriptively compare the outcomes of patients treated on this protocol to a comparable patient population conditioned with whole-body radiotherapy. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of intensity-modulated radiation therapy followed by a phase II study.

PREPARATIVE CHEMOTHERAPY: Patients receive busulfan IV once daily over 2 hours on days -15 and -13 and then every 6 hours on days -12 to -9. Patients also receive etoposide IV on day -3. Patients undergo image-guided intensity-modulated radiation therapy using helical tomotherapy on days -8 to -5.

TRANSPLANTATION: Patients undergo allogeneic peripheral blood stem cell transplantation or bone marrow transplantation on day 0.

GRAFT-VS-HOST DISEASE (GVHD) PROPHYLAXIS: Patients receive GVHD prophylaxis that excludes methotrexate.

After completion of study treatment, patients are followed periodically for 1 year and then annually for 2 years thereafter.

ELIGIBILITY:
Inclusion

* Patients with the following diagnoses are eligible for this study: Advanced myeloid malignancy with a disease status of more than second remission, induction failure, or relapse; Chronic myeloid leukemia in blast crisis; Myelodysplasia, specifically refractory anemia with excess blasts (RAEB)
* All candidates for this study must have a HLA (-A, -B, -C, -DR) identical sibling who is willing to donate bone marrow or primed blood stem cells or a 10/10 allele-matched unrelated donor or minor mismatches as per BMT SOP that allows Tacrolimus and Sirolimus to be given for GVH prophylaxis; all ABO blood group combinations of the donor/recipient are acceptable since even major ABO compatibilities can be dealt with by various techniques (red cell exchange or plasma exchange)
* Prior therapy with VP-16, busulfan, hydrea and gleevec are allowed
* A cardiac evaluation with electrocardiogram and MUGA or echocardiogram is required for all patients; patients must have an ejection fracture of greater than or equal to 50%
* Patients must have a serum creatinine of less than or equal to 1.2 or creatinine clearance > 80 ml/min
* A bilirubin of less than or equal to 1.5; patients should also have an SGOT and SGPT less than 5 times the upper limit of normal
* Pulmonary function tests including DLCO will be performed; FEV1 and DLCO should be greater than 50% of predicted normal value
* Time from the end of last induction or reinduction attempt should be greater than or equal to 21 days
* A signed (IRB approved) informed consent document is required; the patient, donor family member, and transplant team (physician, nurse, and social worker) meet together at least once prior to starting the transplant procedure to review all pertinent risk/benefit information as part of the consenting process; alternative treatment modalities are also discussed at this meeting

Exclusion

* Prior radiation therapy/exposure that prevents patient from receiving IMRT (Determination will be made by the Radiation Oncologist)
* Patients who have previously undergone a blood/marrow transplant and now have relapsed disease
* Patients with a psychological or medical condition that the treating physician deems unacceptable to proceed to allogeneic bone marrow transplant
* Pregnancy
* EKG showing ischemic changes or abnormal rhythm and echocardiogram showing ejection fraction < 50 % or abnormal wall motion

Ages: 6 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2007-06-11 (Actual); Primary Completion 2011-05-17 (Actual); Study Completion 2011-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Stein, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope, Duarte, California, United States

IPD SHARING:
Plan to Share IPD: No
Terminated study

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I: 1200cGy: 1200cGy = 150cGy x 8 doses: Patients receive busulfan IV once daily over 2 hours on days -15 and -13 and then every 6 hours on days -12 to -9. Patients also receive etoposide IV on day -3. Patients undergo image-guided intensity-modulated radiation therapy using helical tomotherapy on days -8 to -5.
  TRANSPLANTATION: Patients undergo allogeneic peripheral blood stem cell transplantation or bone marrow transplantation on day 0.
  GRAFT-VS-HOST DISEASE (GVHD) PROPHYLAXIS: Patients receive GVHD prophylaxis that excludes methotrexate.
  busulfan: Given IV
  etoposide: Given IV
  intensity-modulated radiation therapy: Initially 150 cGy X 8 doses with gradual dose escalation to 200 cGy X 10 doses
  allogeneic hematopoietic stem cell transplantation: Stem cell transplantation occurs on Day 0 after High Dose Therapy
  allogeneic bone marrow transplantation: Stem cell transplantation occurs on Day 0 after High Dose Therapy
  peripheral blood stem cell transplantation: Stem cell transplantation occurs on Day 0 after High Dose Therapy
  tomotherapy: Initially 150 cGy X 8 doses with gradual dose escalation to 200 cGy X 10 doses
Period: Overall Study
Arm/Group | Arm I: 1200cGy | Arm II: 1350cGy
Started | 23 | 2
Completed | 23 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I: 1200cGy | Arm II: 1350cGy | Total
Number analyzed (Participants) | 23 | 2 | 25
Age, Continuous [Median (Full Range); unit: years] | 40 [18 to 56] | 36 [29 to 43] | 40 [18 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 1 | 10
  Male | 14 | 1 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 6
  Not Hispanic or Latino | 17 | 1 | 18
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 0 | 1
  White | 19 | 2 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 23 | 2 | 25

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Intensity-modulated Radiation Therapy (Phase I)
Description: The highest dose tested in which fewer than 33% of patients experienced DLT attributable to the study treatment when at least six patients were treated at the dose and are evaluable for toxicity. The MDT is one dose level below the DLT level. At least six patients will be treated at the MTD.
Time Frame: from initial treatment date to Day 30 post-transplant
Population: 6 patients treated at dose level one (1200cGy) are evaluable for dose limiting evaluable in Phase I.
Measure: Number; unit: cGy
Arm/Group | Arm I: 1200cGy
Number analyzed (Participants) | 6
cGy | 1200

ADVERSE EVENTS:
Time Frame: Adverse events were captured from initial treatment to Day 180 post-transplant. Vital Statuses were captured from the initial treatment to death.
Arm/Group | Arm I: 1200cGy | Arm II: 1350cGy
All-Cause Mortality (participants affected / at risk) | 19/23 | 2/2
Serious Adverse Events (participants affected / at risk) | 7/23 | 2/2
Other Adverse Events (participants affected / at risk) | 23/23 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: 1200cGy (N=23) | Arm II: 1350cGy (N=2)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Ascites (non-malignant) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus, GI (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis/stomatitis (clinical exam) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 (1) | 0 (0)
Febrile neutropenia (ANC <1.0 x 10e9/L, fever >=38.5 degrees C) (Infections and infestations) | 1 (1) | 0 (0)
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) (Infections and infestations) | 2 (2) | 0 (0)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Syndromes - Other (Specify, __) (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: 1200cGy (N=23) | Arm II: 1350cGy (N=2)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 4 (4) | 1 (1)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 4 (4) | 0 (0)
Veno-Occlusive Disease (VOD) (Investigations) | 0 (0) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 22 (22) | 1 (1)
Hemolysis (e.g., immune hemolytic anemia, drug-related hemolysis) (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Iron overload (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 21 (21) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 22 (22) | 2 (2)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 20 (20) | 2 (2)
Platelets (Blood and lymphatic system disorders) | 22 (22) | 2 (2)
Transfusion: Platelets for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Transfusion: pRBCs for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 22 (22) | 2 (2)
Hypertension (Cardiac disorders) | 9 (9) | 1 (1)
Hypotension (Cardiac disorders) | 8 (8) | 2 (2)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (non-malignant) (Cardiac disorders) | 2 (2) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Restrictive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Valvular heart disease (Cardiac disorders) | 1 (1) | 0 (0)
INR (International Normalized Ratio of prothrombin time) (Vascular disorders) | 1 (1) | 0 (0)
PTT (Partial Thromboplastin Time) (Vascular disorders) | 6 (6) | 2 (2)
Thrombotic microangiopathy (Vascular disorders) | 1 (1) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 23 (23) | 2 (2)
Fever (in the absence of neutropenia, ANC <1.0 x 10e9/L) (General disorders) | 8 (8) | 0 (0)
Insomnia (General disorders) | 18 (18) | 0 (0)
Rigors/chills (General disorders) | 16 (16) | 2 (2)
Sweating (diaphoresis) (General disorders) | 2 (2) | 0 (0)
Weight gain (General disorders) | 11 (11) | 1 (1)
Weight gain (General disorders) | 0 (0) | 1 (1)
Weight loss (General disorders) | 10 (10) | 0 (0)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 14 (14) | 1 (1)
Flushing (Skin and subcutaneous tissue disorders) | 14 (14) | 2 (2)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 19 (19) | 2 (2)
Hypopigmentation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Induration/fibrosis (skin and subcutaneous tissue) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 8 (8) | 2 (2)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 8 (8) | 1 (1)
Rash/dermatitis associated with high-dose chemotherapy or BMT studies. (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 22 (22) | 2 (2)
Rash: dermatitis associated with radiation (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 11 (11) | 0 (0)
Ulceration (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Anorexia (Gastrointestinal disorders) | 16 (16) | 1 (1)
Ascites (non-malignant) (Gastrointestinal disorders) | 2 (2) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 8 (8) | 2 (2)
Dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 19 (19) | 2 (2)
Distension/bloating, abdominal (Gastrointestinal disorders) | 13 (13) | 2 (2)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 3 (3) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 4 (4) | 0 (0)
Flatulence (Gastrointestinal disorders) | 5 (5) | 1 (1)
Gastrointestinal - Other (Specify, __) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Heartburn/dyspepsia (Gastrointestinal disorders) | 12 (12) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 6 (6) | 1 (1)
Ileus, GI (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Incontinence, anal (Gastrointestinal disorders) | 3 (3) | 0 (0)
Mucositis/stomatitis (clinical exam) (Gastrointestinal disorders) | 22 (22) | 1 (1)
Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 22 (22) | 1 (1)
Nausea (Gastrointestinal disorders) | 23 (23) | 2 (2)
Proctitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 4 (4) | 0 (0)
Typhlitis (cecal inflammation) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 22 (22) | 2 (2)
Hemorrhage, GI (Vascular disorders) | 9 (9) | 1 (1)
Hemorrhage, GU (Vascular disorders) | 8 (8) | 1 (1)
Hemorrhage, pulmonary/upper respiratory (Vascular disorders) | 9 (9) | 1 (1)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Vascular disorders) | 4 (4) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatobiliary/Pancreas - Other (Specify, __) (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 2 (2) | 0 (0)
Febrile neutropenia (ANC <1.0 x 10e9/L, fever >=38.5 degrees C) (Infections and infestations) | 13 (13) | 1 (1)
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) (Infections and infestations) | 13 (13) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 5 (5) | 1 (1)
Opportunistic infection associated with >=Grade 2 Lymphopenia (Infections and infestations) | 1 (1) | 1 (1)
Infection, Bacterial (COH) (Infections and infestations) | 2 (2) | 0 (0)
Infection, Fungal (COH) (Infections and infestations) | 1 (1) | 0 (0)
Edema:head and neck (General disorders) | 11 (11) | 1 (1)
Edema:limb (General disorders) | 21 (21) | 2 (2)
Edema:trunk/genital (General disorders) | 7 (7) | 0 (0)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 16 (16) | 1 (1)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 20 (20) | 2 (2)
Acidosis (metabolic or respiratory) (Investigations) | 0 (0) | 1 (1)
Albumin, serum-low (hypoalbuminemia) (Investigations) | 21 (21) | 2 (2)
Alkaline phosphatase (Investigations) | 20 (20) | 2 (2)
Alkalosis (metabolic or respiratory) (Investigations) | 3 (3) | 0 (0)
Bicarbonate, serum-low (Investigations) | 15 (15) | 1 (1)
Bilirubin (hyperbilirubinemia) (Investigations) | 9 (9) | 2 (2)
CPK (creatine phosphokinase) (Investigations) | 1 (1) | 0 (0)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 6 (6) | 0 (0)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 21 (21) | 2 (2)
Cholesterol, serum-high (hypercholesteremia) (Metabolism and nutrition disorders) | 5 (5) | 0 (0)
Creatinine (Metabolism and nutrition disorders) | 7 (7) | 2 (2)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 21 (21) | 2 (2)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 7 (7) | 2 (2)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 21 (21) | 2 (2)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 19 (19) | 2 (2)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 6 (6) | 1 (1)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 21 (21) | 2 (2)
Proteinuria (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 7 (7) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 22 (22) | 2 (2)
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 20 (20) | 1 (1)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 5 (5) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 13 (13) | 1 (1)
Musculoskeletal/Soft Tissue - Other (Specify, __) (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Confusion (Nervous system disorders) | 9 (9) | 2 (2)
Dizziness (Nervous system disorders) | 4 (4) | 0 (0)
Mood alteration (Nervous system disorders) | 21 (21) | 2 (2)
Neuropathy: cranial (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy: motor (Nervous system disorders) | 2 (2) | 0 (0)
Neuropathy: sensory (Nervous system disorders) | 3 (3) | 1 (1)
Somnolence/depressed level of consciousness (Nervous system disorders) | 4 (4) | 0 (0)
Tremor (Nervous system disorders) | 6 (6) | 0 (0)
Dry eye syndrome (Eye disorders) | 8 (8) | 1 (1)
Ocular/Visual - Other (Specify, __) (Eye disorders) | 1 (1) | 0 (0)
Vision-blurred vision (Eye disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 23 (23) | 2 (2)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 2 (2)
FEV(1) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 1 (1)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Cystitis (Renal and urinary disorders) | 1 (1) | 0 (0)
Incontinence, urinary (Renal and urinary disorders) | 3 (3) | 1 (1)
Renal failure (Renal and urinary disorders) | 5 (5) | 0 (0)
Renal/Genitourinary - Other (Specify, __) (Renal and urinary disorders) | 2 (2) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1 (1) | 0 (0)
Urine color change (Renal and urinary disorders) | 3 (3) | 0 (0)
Vaginal discharge (non-infectious) (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginitis (not due to infection) (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Syndromes - Other (Specify, __) (Investigations) | 4 (4) | 0 (0)
Tumor lysis syndrome (Investigations) | 1 (1) | 0 (0)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 4 (4) | 0 (0)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-06-29): https://cdn.clinicaltrials.gov/large-docs/95/NCT00540995/Prot_SAP_000.pdf